CLINICAL TRIAL: NCT06049888
Title: Causal Effects of Exposure to Social Media on Adolescent Mental Health
Brief Title: Does Social Media Impact Adolescent Mental Health?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 1R01MH135467 (NIH)
Record Dates: First submitted 2023-08-23; First posted 2023-09-22 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Mental Health
Keywords: social media; mental health; depression; anxiety
MeSH Terms: conditions — Psychological Well-Being; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naturalistic Social Media (No Intervention): In this control condition, participants will have no study-imposed restrictions on social media use.
- Restricted Social Media (Experimental): Participants will have social media apps on their phones blocked for three months.
  Interventions: Behavioral: Restricted Social Media

INTERVENTIONS:
Behavioral: Restricted Social Media — Participants (N = 500) will be randomly assigned to either have no study-imposed restrictions on social media use (naturalistic social media condition) or have no access to social media apps on their phones (restricted social media condition). This manipulation will last three months, after which both groups will have no study-imposed restrictions on social media for three more months.
  Arms: Restricted Social Media

SUMMARY:
The mental health of adolescents in the United States has seen a steep decline since 2011, roughly coinciding with the increasing popularity of social media and smartphones. But does social media have a causal impact on the mental health of adolescents or are concerns about the effect of social media on kids a form of public hysteria? In this study, the investigators will conduct the first field experiment in 11-14-year-olds to examine whether, how, and for whom social media harms mental health.

ELIGIBILITY:
Inclusion Criteria:

1. is an adolescent who is between the ages of 10 and 14;
2. is an adolescent whose parents have decided to buy them their first smartphone;
3. is an adolescent both of whose parents/guardians consent for them to be in the study;
4. is an adolescent who assents to be in the study; 5) is an adolescent who speaks and reads English sufficiently to complete surveys and provide informed consent.

Exclusion Criteria:

1. is an adolescent who has severe developmental problems (e.g., autism, severe language delay);
2. is an adolescent who is currently or has ever been diagnosed with severe or moderately severe mental illness;
3. is an adolescent who is currently or has ever experienced suicidal ideation.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2024-09-29 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Revised Child Anxiety and Depression Scale (RCADS-25): Total Score | Baseline, three months, and six months
  The average score varies between 0 and 4, with higher scores indicating a worse outcome.

SECONDARY OUTCOMES:
Revised Child Anxiety and Depression Scale (RCADS-25): Depression Subscale | Baseline, three months, and six months
  The average score varies between 0 and 4, with higher scores indicating a worse outcome.
Revised Child Anxiety and Depression Scale (RCADS-25): Anxiety Subscale | Baseline, three months, and six months
  The average score varies between 0 and 4, with higher scores indicating a worse outcome.

OTHER OUTCOMES:
DSM-5 Self-Rated Level 1 Cross-Cutting Symptom Measure Youth Self Report | Baseline, three months, and six months
  The average score varies between 0 and 4, with higher scores indicating a worse outcome.
DSM-5 Self-Rated Level 1 Cross-Cutting Symptom Measure Parent Report | Baseline, three months, and six months
  The average score varies between 0 and 4, with higher scores indicating a worse outcome.
Upward Social Comparison (EMA) | Every three days throughout the study with two averages computed for 0 to 3 months and 3 to 6 months.
  Mediator measured with a single, face-valid item in EMA surveys: "Over the past 24 hours, how often have you compared yourself to someone who you believe is better off than you?"
Offline Social Capital: Quantity of In-Person Social Interactions (EMA) | Every three days throughout the study with two averages computed for 0 to 3 months and 3 to 6 months.
  Mediator measured with a single, face-valid item in EMA surveys: "Over past 24 hours, how much time did you spend socializing in person?"
Offline Social Capital: Quality of In-Person Social Interactions (EMA) | Every three days throughout the study with two averages computed for 0 to 3 months and 3 to 6 months.
  Mediator measured with a single, face-valid item in EMA surveys: "Over past 24 hours, how much did you enjoy your in-person social interactions with others?"
Quantity of Online Social Interactions (Mobile Sensing) | Daily throughout the study with two averages computed for 0 to 3 months and 3 to 6 months.
  Mediator: Quantity of digital social interactions based on the total number of words participants type on their phone keyboards each day.
Valence of Online Social Interactions (Mobile Sensing) | Daily throughout the study with two averages computed for 0 to 3 months and 3 to 6 months.
  Mediator: Quality/valence of digital social interactions by measuring the balance between positive and negative words participants type on their phone keyboards. The valence of the words typed will first be scored using the Linguistic Inquiry and Word Count (LIWC) software. The sum of the valence scores of all words will produce the final score for analysis.
Active (vs Passive) Social Media Use (Mobile Sensing) | Daily throughout the study with two averages computed for 0 to 3 months and 3 to 6 months.
  Active usage includes creating content and direct messaging, while passive usage includes browsing, scrolling, or watching videos. Using data from the Inertial Measurement Unit (i.e., accelerometer and gyroscope data) and keyboard input (i.e. typing or not), an Extremely Randomized Trees algorithm will classify behaviors into active or passive.
Passive (vs Active) Social Media Use (Mobile Sensing) | Daily throughout the study with two averages computed for 0 to 3 months and 3 to 6 months.
  Active usage includes creating content and direct messaging, while passive usage includes browsing, scrolling, or watching videos. Using data from the Inertial Measurement Unit (i.e., accelerometer and gyroscope data) and keyboard input (i.e. typing or not), an Extremely Randomized Trees algorithm will classify behaviors into active or passive.
Time Spent in Specific Social Media Apps (Mobile Sensing) | Daily throughout the study with two averages computed for 0 to 3 months and 3 to 6 months.
  Time participants spend in specific social media apps as assessed unobtrusively by mobile sensing.

CONTACTS AND LOCATIONS:
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
Demographic, clinical (self-reports and parent reports), neurocognitive (gradCPT), and passive mobile sensing data (accelerometer, GPS, keyboard input, app usage) will be collected and made available on NIMH Data Archive (NDA). All data will be de-identified prior to deposition to NDA. To request access to the data, researchers will use the standard processes at NDA, and the NDA Data Access Committee will decide which requests to grant. All code for the analyses-including statistical analysis, data transformations, and data cleaning-will be shared on the Open Science Framework (OSF). The code can be found by searching for "Kostadin Kushlev" on the Open Science Framework.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: All data will be deposited to NDA starting 12 months after the award begins and will be deposited every six months thereafter following the usual NDA data submission dates.
Access Criteria: To request access to the data, researchers will use the standard processes at NDA, and the NDA Data Access Committee will decide which requests to grant. The standard NDA data access process allows access for one year and is renewable. The protocol and code will be available on OSF to anybody with access to the internet. De-identified data associated with each publication will also be made available on OSF by the publication date of each paper.